CLINICAL TRIAL: NCT04283331
Title: Efficacy and Safety of Anesthetic Impregnated Bandage Soft Contact Lens (BSCL) in Pain Management After Photorefractive Keratectomy (PRK).
Brief Title: Anesthetic Impregnated Bandage Soft Contact Lens (BSCL) in Pain Management After Photorefractive Keratectomy (PRK)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beeran Meghpara, MD (Other)
Responsible Party: Sponsor-Investigator, Beeran Meghpara, MD, Clinical Assistant Professor of Ophthalmology, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 19-871
Record Dates: First submitted 2020-02-16; First posted 2020-02-25 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Myopia; Hypermetropia; Refractive Errors; Astigmatism
Keywords: refractive surgery; PRK; LASIK
MeSH Terms: conditions — Myopia; Hyperopia; Refractive Errors; Astigmatism | interventions — proxymetacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The laser vision technician will be the only member aware of which eye received the control vs intervention treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bandage Contact Lens + Proparacaine (Experimental): The eye that receives a bandage contact lens soaked in proparacaine.
  Interventions: Drug: Proparacaine Ophthalmic
- Bandage Contact Lens WITHOUT Proparacaine (No Intervention): The eye that receives a bandage contact lens (standard of care).

INTERVENTIONS:
Drug: Proparacaine Ophthalmic — Each subject will have one eye randomized to receive a bandage contact lens soaked in anesthetic solution (proparacaine hydrochloride 0.5%) and the following eye will serve as a control and receive a bandage soft contact lens soaked in balanced salt solution, which is the current standard of care for PRK.
  Other Names: Proparacaine; proparacaine hydrochloride 0.5%
  Arms: Bandage Contact Lens + Proparacaine

SUMMARY:
Compared to laser-assisted in situ keratomileusis (LASIK), Photorefractive Keratectomy (PRK) is associated with more discomfort and requires more downtime. However, it is oftentimes considered the preferred method of refractive surgery for patients with dry eye syndrome, high refractive errors, thin corneas, or those with more active lifestyles who may be more prone to dislodging their LASIK flaps. We hypothesize that the use of bandage contact lenses soaked in proparacaine will decrease pain levels compared to solely the use of bandage contact lenses after PRK.

DETAILED DESCRIPTION:
Photorefractive keratectomy (PRK) is a popular method for the correction of refractive errors. Compared to laser-assisted in situ keratomileusis (LASIK), PRK is often associated with more discomfort and requires more downtime. However, it is oftentimes considered the preferred method of refractive surgery for patients with dry eye syndrome, high refractive errors, thin corneas, or those with more active lifestyles who may be more prone to dislodging their LASIK flaps. It can also avoid other complications associated with LASIK including striae, folds, diffuse lamellar keratitis, and epithelial ingrowth. As a result, improved management of post-operative pain in patients undergoing PRK is critical in order encourage utilization and patient preference of this procedure.

The current standard of care for pain management after PRK is the use of a bandage soft contact lens (BSCL). BSCLs may speed reepithelialization and function as an adjunct for pain control.

Using a BSCL soaked in proparacaine has not yet been studied as a pain management method after PRK. Our hypothesis is that combining these two methods will result in greater pain reduction than using a BSCL alone, which is the current standard of care. Furthermore, soaking the BSCL in anesthetics will reduce the chance that patients can abuse anesthetic medication postoperatively, which is the concern when patients are sent home with anesthetic drops as is noted in several prior studies.

This study aims to explore the potential of an anesthetic soaked bandage soft contact lens in reducing pain levels compared to a bandage soft contact lens alone after PRK.

Study Goals:

* To assess the perception of pain following photorefractive keratectomy with the utilization of an anesthetic soaked bandage soft contact lens versus control (BSCL only) using the Visual Analog Pain Scale.
* To assess the effect of an anesthetic soaked bandage soft contact lens on re-epithelialization following photorefractive keratectomy versus control. This will be assessed on post-operative day 5 as whether there is a persistent epithelial defect or not, a binary outcome.

ELIGIBILITY:
Inclusion Criteria:

* All eyes approved for photorefractive keratectomy with Dr. Beeran Meghpara or Dr. Christopher Rapuano, with or without the assistance of residents.

Exclusion Criteria:

* Patients undergoing unilateral procedure.
* Eyes that experience complication during the photorefractive keratectomy procedure
* Patients who are pregnant or breast feeding
* Patients under 18 years of age
* Patients with a history of eye surgery or trauma and those with irregular astigmatism, keratoconus, or any other type of corneal disorder, pregnancy, diabetic retinopathy, or glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily pain score at post-operative day 0 through post-operative day 5 | 5 days
  Primary Outcome Measure is pain score at post-operative day 0 THROUGH post-operative day 5. Patients will be asked to fill out their score daily.
  The Wong-Baker Faces pain scale will be used to measure pain. This is a self-report measure of pain consisting of a series of faces with expressions of increasing distress. Each face is also given a numerical rating from 0 to 5, zero representing no pain and 5 representing worst pain.

SECONDARY OUTCOMES:
Complete re-epithelialization at post-operative day 5 | 5 days
  A binary outcome (yes/no) of whether the corneal epithelium has completely healed by post-operative day 5.
Final refractive outcome at postoperative month 3 | 3 Months
  Snellen visual acuity, both without correction and best corrected with a manifest refraction.

CONTACTS AND LOCATIONS:
Overall Officials: Beeran Meghpara, MD, Principal Investigator — Wills Eye Hospital at TJUH
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States